CLINICAL TRIAL: NCT01647477
Title: Determinants of the Consultation Delay in Cancers of the Upper Aero Digestive Tract
Brief Title: Interventional Study Collecting Quantitative and Qualitative Data About Patient With Non Treated Cancer
Acronym: DEREDIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEREDIA - 1110
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Upper Aerodigestive Tract Cancer
Keywords: non treated cancer; oral cavity; oropharynx; hypopharynx; larynx; first consultation
MeSH Terms: conditions — Laryngeal Diseases | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- questionnaires (Active Comparator): 4 questionnaires to answer at baseline 45 minutes approx.
  Interventions: Behavioral: questionnaires
- interview (Experimental): semi directive interview 105 patients
  Interventions: Behavioral: interview; Behavioral: questionnaires

INTERVENTIONS:
Behavioral: interview — 25 minutes of semi directive interview
  Arms: interview
Behavioral: questionnaires — questionnaires to answer at baseline 45 minutes

SUMMARY:
This study aims to determine the impact of sociocognitive and emotional factors on the time of the initial consult

DETAILED DESCRIPTION:
identify wich sociocognitive factors influence the delay to go to a doctor after the emergence of first symptoms

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* oral cavity cancer, oropharynx cancer, hypopharynx cancer, larynx cancer
* non treated cancer
* patient informed of his diagnosis
* speak fluent french
* patient covered by health insurance
* signed informed consent

Inclusion Criteria for "interviewed " patients :

* no speech troubles
* patient consents being recorded

Exclusion Criteria:

* history of cancer
* psychological history
* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
time of first consultation | baseline
  median time between date of symptoms appearance and date of first consultation

SECONDARY OUTCOMES:
identify variables associated with time of consultation | baseline
  medical data : medical history, symptoms, entry into care pathway sociodemographic and emotional indicators

CONTACTS AND LOCATIONS:
Overall Officials: Veronique CHRISTOPHE, MDPhD, Study Director — Lille 3 University
Locations (7):
- France (7):
  - Centre Hospitalier, Boulogne-sur-Mer
  - CH, Lens
  - Oscar Lambret Center, Lille
  - Centre Hospitalier Régional et Universitaire - Hopital HURIEZ, Lille
  - La Louviere Hospital, Lille
  - Gray Center, Maubeuge
  - Centre Médical Spécialisé du Littoral, Saint Martin Les Boulogne

IPD SHARING:
Plan to Share IPD: No